CLINICAL TRIAL: NCT00762606
Title: A Twelve-Months, Single-Masked, Parallel Group, Health Economic Study of Phacoemulsification Versus Small Incision Cataract Surgery (SICS) in Chinese Patients With Senile Cataract.
Brief Title: Phaco Versus Small Incision Cataract Surgery (SICS) Health Economic Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RM-08-002
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Results first posted 2011-07-08 (Estimated); Last update posted 2012-10-31 (Estimated); Status verified 2011-08

CONDITIONS: Cataract
Keywords: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phaco (Active Comparator): Cataract extraction surgery utilizing Phacoemulsification
  Interventions: Procedure: Phacoemulsification cataract extraction surgery
- SICS (Active Comparator): Small incision cataract surgery (SICS)
  Interventions: Procedure: Small incision cataract surgery

INTERVENTIONS:
Procedure: Phacoemulsification cataract extraction surgery — Surgical removal of cataract using phacoemulsification followed by implantation of an AcrySof Intraocular Lens (Model SN60WF)
  Arms: Phaco
Procedure: Small incision cataract surgery — Surgical removal of cataract using small incision cataract surgery (SICS) followed by implantation of a Polymethyl methacrylate(PMMA) Intraocular Lens (Model MZ60BD).
  Arms: SICS

SUMMARY:
To compare the health economic parameter and clinical outcome of Phacoemulsification with small incision cataract surgery (SICS)

ELIGIBILITY:
Inclusion Criteria:

* Patient has senile cataract and require unilateral cataract extraction followed by implantation of an AcrySof or PMMA (polymethylmethacrylate) posterior chamber intraocular lens (IOL);
* Pupil dilation ≧7 mm after mydrisis;
* Patient undergoing cataract surgery for the first eye;
* VA prognosis ≧6/12

Exclusion Criteria:

* Patients with history of ocular pathology or diabetic retinopathy;
* Patients with traumatic, subluxated and posterior polar cataract;
* Patients had ocular surgery in the past 6 months;
* Patients with significant intra-operative complications

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2008-09; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Alcon Call Center, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Phaco | SICS
Started | 55 | 51
Completed | 37 | 38
Not Completed | 18 | 13
Not completed — Lost to Follow-up | 18 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phaco | SICS | Total
Number analyzed (Participants) | 55 | 51 | 106
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 11 | 19
  >=65 years | 47 | 40 | 87
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 31 | 64
  Male | 22 | 20 | 42

OUTCOME MEASURES:

1. Primary Outcome: Posterior Capsule Opacification Evaluation
Description: The number of subjects with Posterior Capsular Opacification (PCO) for 12 months post-surgery of the study eye. PCO may occur after cataract surgery and is caused by residual lens epithelial cells that remain in the capsular bag after surgery and undergo proliferation, migration, and fibrous metaplasia. PCO was evaluated via slit lamp. A lower PCO rate is better.
Time Frame: 12 months after surgery
Measure: Number; unit: participants
Arm/Group | Phaco | SICS
Number analyzed (Participants) | 36 | 38
participants | 3 | 28

2. Secondary Outcome: Corneal Astigmatism
Description: Analysis of corneal astigmatism 12 months after surgery using Orbscan Topography. A lower corneal astigmatism value is better.
Time Frame: 3 months after surgery
Measure: Mean (Standard Deviation); unit: Diopters
Arm/Group | Phaco | SICS
Number analyzed (Participants) | 55 | 51
Diopters | 1.05 (0.80) | 1.95 (1.15)

ADVERSE EVENTS:
Time Frame: During surgery, 1 day,2 weeks, 1 month, 3 months,6 months and 12 months after surgery.
Arm/Group | Phaco | SICS
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/51
Other Adverse Events (participants affected / at risk) | 2/55 | 6/51
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phaco (N=55) | SICS (N=51)
Posterior Capsular Rupture (Eye disorders) | 2 (2) | 3 (3)
Conjunctival Congestion (Eye disorders) | 0 (0) | 1 (1)
Femoral Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Zonular Rupture (Eye disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No